CLINICAL TRIAL: NCT03114761
Title: Abdominal CT Angiography of Mesenteric Vessels for Diagnosing Internal Herniation After Roux-en-Y Gastric Bypass Surgery
Brief Title: CTA for Internal Herniation After RYGB Surgery
Acronym: CTA-IH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Laura Deden, Principal Investigator, Rijnstate Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL52257.091.15
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Internal Hernia
Keywords: Roux-en-Y Gastric Bypass; Internal Herniation; Computed Tomography
MeSH Terms: conditions — Internal Hernia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CTA-IH (Experimental)
  Interventions: Radiation: CT angiography

INTERVENTIONS:
Radiation: CT angiography — Patients are subjected to a standard abdominal CT scan and (additional in this study) to abdominal CT angiography (CTA)

SUMMARY:
Introduction: Morbid obesity, defined as a body mass index (BMI) of over 40 kg/m2, is globally an imminent health threat. Conservative therapies do often not yield the desired result. Bariatric surgery includes several interventions that are performed on patients with morbid obesity, like gastric bypass surgery. The number of bariatric surgeries annually is estimated to be around 500,000 worldwide; about half of these are gastric bypass surgeries. In the Netherlands, the most common performed bariatric intervention is the Roux-en-Y gastric bypass (RYGB). An important long-term complication of this surgery is internal herniation, a condition in which a part of the GI tract is herniated through an opening in the mesentery made during RYGB surgery. Incidence of internal herniation is 1-5%. Conventional abdominal CT examination is often not conclusive about the presence of internal herniation. When internal herniation is clinically highly suspected after abdominal CT examination (but not necessarily confirmed), the patient is subjected to diagnostic laparoscopic surgery. Unfortunately, a negative abdominal CT scan does not exclude internal herniation in all patients. This pleads for the development or exploitation of alternative techniques that might aid in the diagnosis of complications after RYGB surgery. Since the anatomy of GI tract is altered when internal herniation is present, visualizing the mesenteric vasculature may aid in the diagnosis of this complication after RYGB surgery. This study aims to confirm the feasibility and superiority of diagnosing internal herniation using CT examination of the mesenteric arteries over conventional CT examination.

Objectives: The primary objective is to determine whether abdominal arterial CT angiography is a feasible technique for diagnosing internal herniation after RYGB surgery. Secondary, it is examined whether arterial angiography of the mesentery is superior over conventional CT examination with oral and IV contrast in the venous phase.

Study design: This study will be a prospective pilot study, in which the outcomes of both the conventional CT examination and abdominal angiogram are compared to the outcome of diagnostic laparoscopy as gold standard.

Study population: Patients will be included who underwent laparoscopic RYGB surgery at least half a year earlier and have persisting abdominal pain. They should be highly suspected for internal herniation by their doctor, based on several characteristics.

Main study parameters/endpoints: Primary study endpoints are the assessments of the arterial abdominal angiogram and mesenteric arterial mapping in relation to the outcome of the diagnostic laparoscopic surgery in 12 subjects.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In this pilot study, study subjects will receive an additional effective radiation dose of about 10 mSv. On average, an acute dose of 10 mSv leads to an additional risk of cancer of about 1 in 1750 (~1 in 2000 for males, ~1 in 1500 for females) for a 50-year old subject, based on the linear no threshold model. However, when the mesenteric artery mapping proves to be feasible and superior, many unnecessary diagnostic laparoscopic surgeries will be prevented (along with their complications and risks).

ELIGIBILITY:
Inclusion Criteria:

* The patient should have underwent laparoscopic RYGB surgery (standard procedure with closing of mesenteric openings) at least half a year earlier;
* The patient should have abdominal pain, at least three days in a row;
* The patient should be highly suspected for internal herniation by their doctor (based on weight loss, location of pain, intervals between pain, relation to food intake).

Exclusion Criteria:

* The patient has an age below 18;
* The patient is incompetent to decide;
* The patient is pregnant or gives breast feeding;
* The patient is in emergency setting and requires imminent surgery;
* The patient has other known abdominal pathology or prior large abdominal surgery;
* The patient has had surgery for internal herniation previously;
* The patient has had earlier surgery involving the RYGB, such as distalisation;
* One or both scans have insufficient scan quality;
* The patient will not be subjected to diagnostic laparoscopic surgery (e.g. pain-free patients);
* The patient has a contra-indication for the administration of oral or IV contrast (Xenetide 300mg/ml).:

  * Thyrotoxicose
  * Overgevoeligheid/allergisch voor Xenetix of in het verleden een allergische reactie op jodiumhoudend contrast
  * Treatment with NSAID's, diuretica or aminoglycosiden that cannot be stopped 24 hours before and after the CT
  * Treatment with cisplatina less than six weeks before CT
  * M.Kahler or M. Waldenstrom
  * Kidneyfunction (GFS) < 60

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
CTA examination | 1 year
  Assessment of the CT-angiography for the presence of internal herniation and comparing outcome to laparoscopic evalutation (gold standard)

SECONDARY OUTCOMES:
Standard CT examination | 1 year
  Standard radiologic examination of the standard CT, i.e. for the presence of internal herniation and comparison to the findings on CT-angiography and laparascopy

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate hospital, Arnhem, Netherlands